CLINICAL TRIAL: NCT01562379
Title: Evaluation of Complementary Food Supplements For Reducing Childhood Undernutrition: The JiVitA-4 Study
Brief Title: Complementary Food Supplements for Reducing Childhood Undernutrition
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); United Nations World Food Programme (WFP) (Other); DSM Ltd (Industry)
Responsible Party: Principal Investigator, Parul Christian, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00003703; NIFA210-38418-21732 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2012-03-09; First posted 2012-03-23 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-12

CONDITIONS: Stunting; Wasting
Keywords: complementary food supplements; stunting; wasting; growth; Bangladesh; infant feeding
MeSH Terms: conditions — Growth Disorders; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- No food (No Intervention): A control in which mothers will receive nutrition education about continued breastfeeding and adequate complementary feeding throughout the period of 6-18 months of age.
- Plumpy Doz (Active Comparator): In this control arm children will receive prepackaged, lipid-based Plumpy'Doz (Nutriset, Mulaunay, France) for daily consumption as a snack.
  Interventions: Dietary Supplement: Plumpy Doz
- Wheat Soy Blend (WSB++) (Experimental): Children will receive a WFP-developed Wheat-Soy Blend (WSB++) snack to be consumed daily.
  Interventions: Dietary Supplement: Wheat Soy Blend (WSB++)
- Chickpea based complementary food supplement (Experimental): Children will receive a Chickpea based complementary food supplement to be consumed daily.
  Interventions: Dietary Supplement: Chickpea based complementary food supplement
- Rice based complementary food supplement (Experimental): Children will receive a locally developed rice based complementary food supplement.
  Interventions: Dietary Supplement: Rice based complementary food supplement

INTERVENTIONS:
Dietary Supplement: Wheat Soy Blend (WSB++) — A wheat formulation containing protein from milk solids and soybeans, essential fats and sugar to provide optimal caloric density, and added vitamins and minerals.
  Arms: Wheat Soy Blend (WSB++)
Dietary Supplement: Chickpea based complementary food supplement — A chickpea-based complementary food supplement with added milk powder, oil, sugar and added vitamins and minerals.
  Arms: Chickpea based complementary food supplement
Dietary Supplement: Rice based complementary food supplement — Locally developed rice based complementary food with and added vitamins and minerals.
  Arms: Rice based complementary food supplement
Dietary Supplement: Plumpy Doz — Plumpy Doz is a prepackaged ready-to-use complementary food supplement enriched with added vitamins and minerals.
  Arms: Plumpy Doz

SUMMARY:
The purpose of this study is to test the impact on child growth of three specially formulated complementary food supplements vs. Plumpy'Doz, a previously tested, commercially available complementary food, and vs. a control group that receives no food. All groups will receive nutrition education related to infant and young child feeding. This will be a cluster-randomised trial in children 6-18 months old in rural Rangpur and Gaibandha in Bangladesh.

DETAILED DESCRIPTION:
Childhood stunting and growth faltering is highly prevalent in South Asia. Among other strategies, adequate complementary feeding practices and provision of complementary foods that are appropriate and fill the nutrient gap by providing macro and micronutrients essential for growth are important means to reduce the global burden of undernutrition and related morbidity and mortality.

We propose to evaluate the impact of three complementary food supplement products that are fortified with micronutrients in a rural, remote setting in Bangladesh, where high rates of childhood undernutrition persist on child growth, health, and development. The three foods being tested are an enhanced wheat-soy blend (WSB++) developed by WFP, and locally developed chickpea-based and a rice-based complementary food supplements.

We will assess the impact of feeding these daily against the non-fed controls, hypothesizing that the children fed these foods show increased length for age Z scores (LAZ) and weight for length age Z scores (WLZ) of >0.21 and decreased prevalence of stunting and wasting by >10%. We expect that the impact of the three foods will be equivalent/ non-inferior to that of Plumpy'Doz.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6 months of age

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5449 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parul Christian, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Keith P West, DrPH, Study Director — Johns Hopkins Bloomberg School of Public Health; Rolf Klemm, DrPH, Study Director — Johns Hopkins Bloomberg School of Public Health; Alain B Labrique, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Kerry J Schulze, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Sucheta Mehra, MS, Study Director — Johns Hopkins Bloomberg School of Public Health; Rebecca Merrill, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Abu Ahmed Shamim, MS, Study Director — JiVitA; Hasmot Ali, MPH, Study Director — JiVitA; Tahmeed Ahmed, PhD, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh; Saskia de Pee, PhD, Study Director — WFP; Martin Bloem, PhD, Study Director — WFP; Monira Parveen, PhD, Study Director — WFP; Britta Schumacher, PhD, Study Director — WFP
Locations (1):
- The JiVitA Project, Johns Hopkins Bangladesh, Gaibandha, Bangladesh

REFERENCES:
- [Derived] Pasqualino MM, Campbell RK, Hurley KM, Wu LS, Shamim AA, Shaikh S, de Pee S, Christian P. Complementary Food Supplements Fill Energy and Protein Gaps among Children with Dietary Inadequacy in a Complementary Feeding Trial in Rural Bangladesh. J Nutr. 2025 Feb;155(2):602-611. doi: 10.1016/j.tjnut.2024.12.001. Epub 2024 Dec 9. PMID 39662676
- [Derived] Chowdhury ZT, Hurley KM, Campbell RK, Shaikh S, Shamim AA, Mehra S, Christian P. Novel Method for Estimating Nutrient Intakes Using a Semistructured 24-Hour Diet Recall for Infants and Young Children in Rural Bangladesh. Curr Dev Nutr. 2020 Jul 15;4(9):nzaa123. doi: 10.1093/cdn/nzaa123. eCollection 2020 Sep. PMID 32875267
- [Derived] Shaikh S, Campbell RK, Mehra S, Kabir A, Schulze KJ, Wu L, Ali H, Shamim AA, West KP, Christian P. Supplementation with Fortified Lipid-Based and Blended Complementary Foods has Variable Impact on Body Composition Among Rural Bangladeshi Children: A Cluster-Randomized Controlled Trial. J Nutr. 2020 Jul 1;150(7):1924-1932. doi: 10.1093/jn/nxaa061. PMID 32240304
- [Derived] Campbell RK, Hurley KM, Shamim AA, Shaikh S, Chowdhury ZT, Mehra S, Wu L, Christian P. Complementary Food Supplements Increase Dietary Nutrient Adequacy and Do Not Replace Home Food Consumption in Children 6-18 Months Old in a Randomized Controlled Trial in Rural Bangladesh. J Nutr. 2018 Sep 1;148(9):1484-1492. doi: 10.1093/jn/nxy136. PMID 30184222
- [Derived] Campbell RK, Schulze KJ, Shaikh S, Mehra S, Ali H, Wu L, Raqib R, Baker S, Labrique A, West KP Jr, Christian P. Biomarkers of Environmental Enteric Dysfunction Among Children in Rural Bangladesh. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):40-46. doi: 10.1097/MPG.0000000000001557. PMID 28644348
- [Derived] Campbell RK, Hurley KM, Shamim AA, Shaikh S, Chowdhury ZT, Mehra S, de Pee S, Ahmed T, West KP Jr, Christian P. Effect of complementary food supplementation on breastfeeding and home diet in rural Bangladeshi children. Am J Clin Nutr. 2016 Nov;104(5):1450-1458. doi: 10.3945/ajcn.116.135509. Epub 2016 Sep 28. PMID 27680994

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Food | Plumpy Doz | Wheat Soy Blend (WSB++) | Chickpea Based Complementary Food Supplement | Rice Based Complementary Food Supplement
Started | 1438 | 1492 | 851 | 843 | 825
Completed | 1312 | 1395 | 789 | 786 | 785
Not Completed | 126 | 97 | 62 | 57 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Food | Plumpy Doz | Wheat Soy Blend (WSB++) | Chickpea Based Complementary Food Supplement | Rice Based Complementary Food Supplement | Total
Number analyzed (Participants) | 1438 | 1492 | 851 | 843 | 825 | 5449
Age, Continuous [Mean (Standard Deviation); unit: months] | 6.13 (0.0) | 6.26 (0.26) | 6.26 (0.27) | 6.24 (0.25) | 6.25 (0.25) | 6.23 (0.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 752 | 725 | 432 | 424 | 425 | 2758
  Male | 686 | 767 | 419 | 419 | 400 | 2691
Region of Enrollment [Number; unit: participants]
  Bangladesh | 1438 | 1492 | 851 | 843 | 852 | 5476

OUTCOME MEASURES:

1. Primary Outcome: Stunting in Children at 18 mo
Description: Prevalence of stunting at 18 months of age.
Time Frame: 18 months of age
Population: Children followed after 1 year of supplementation from 6 months at 18 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | No Food | Plumpy Doz | Wheat Soy Blend (WSB++) | Chickpea Based Complementary Food Supplement | Rice Based Complementary Food Supplement
Number analyzed (Participants) | 1265 | 1344 | 770 | 769 | 755
Participants | 559 | 542 | 341 | 300 | 330

2. Secondary Outcome: Morbidity
Description: weekly morbidity will be assessed for a year and episodes of diarrhea, dysentery ALRI, and fever will be recorded.
Time Frame: weekly from 6 to 18 months of age
Reporting Status: Not Posted

3. Secondary Outcome: Body Composition
Description: Bioelectrical impedance analysis will be used to look at body composition changes from baseline until 18 months of age
Time Frame: At 6, 9 and 12 months of age
Reporting Status: Not Posted

4. Secondary Outcome: Developmental Milestones
Description: Age-specific developmental milestones will be assessed
Time Frame: At 6, 12, and 18 months of age
Reporting Status: Not Posted

5. Secondary Outcome: Cognitive and Motor Function
Description: Using Bayley III
Time Frame: At 18 months of age
Reporting Status: Not Posted

6. Secondary Outcome: Micronutrient Status
Description: Iron, vitamin A, zinc and other micronutrient status of children will be examined by intervention group.
Time Frame: 18 months of age
Reporting Status: Not Posted

7. Secondary Outcome: Intestinal Function
Description: Intestinal function using L:M and other biomarkers will be assessed by intervention group and its association with child growth
Time Frame: At 24 months of age
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Maternal Knowledge, Attitude and Practice Related to Infant and Young Child Feeding
Description: Maternal KAP
Time Frame: At 6, 12 and 18 months of age
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | No Food | Plumpy Doz | Wheat Soy Blend (WSB++) | Chickpea Based Complementary Food Supplement | Rice Based Complementary Food Supplement
All-Cause Mortality (participants affected / at risk) | 12/1438 | 9/1492 | 8/851 | 6/843 | 2/825
Serious Adverse Events (participants affected / at risk) | 0/1438 | 0/1492 | 0/864 | 0/860 | 0/838
Other Adverse Events (participants affected / at risk) | 0/1438 | 0/1492 | 0/851 | 0/843 | 0/825

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No